CLINICAL TRIAL: NCT05831904
Title: Effect of Vibration Therapy on Hip Girdle Muscles in Healthy People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B-2212-801-305
Record Dates: First submitted 2023-04-16; First posted 2023-04-26 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Hip Dislocation
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 20 healthy children (Experimental): 20 healthy children aged 5 to 15 years , without any congenital or developmental abnormalities of their hip joint
  Interventions: Device: whole-body vibration

INTERVENTIONS:
Device: whole-body vibration — After attaching the surface electromyography(EMG) to bilateral hip girdle muscles, participants will walk and jump at their comfortable speed. After investigator record the muscle activation values, participants will be asked to stand on the vibration device. While the whole-body vibration is applied, the hip girdle muscles activation values will be recorded accordingly via sEMG.

SUMMARY:
This clinical trial(prospective, pilot study) is to learn about the effect of whole-body vibration on hip girdle muscles in healthy children as a primary study aiming for a new clinical intervention protocol to prevent hip dislocation in patients with severe cerebral palsy.

DETAILED DESCRIPTION:
Design: Prospective, pilot study Setting: hospital rehabilitation department Intervention: Participants will be asked to walk and jump with a surface electromyography(EMG) attached to their hip girdle muscles. After the participants are positioned(standing) on the platform of whole-body vibration device, the study practitioner will record the sEMG values from the hip girdle muscles during the vibration applied. The mean values of repeating the same process with different vibrations applications and the values before vibration will be compared by using the SPSS using the paired "t-test" or Wilcoxon signed rank test for comparison between before and after vibration in the same group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children (5 to 15 years old)

Exclusion Criteria:

* Children with cerebral palsy, muscle paralysis, developmental or congenital hip joint abnormalities
* Children who underwent hip joint surgery

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
muscle activation values on surface electromyography(sEMG) | 10 seconds for each session
  surface muscle contraction of bilateral hip girdle muscles
  bilateral gluteus medius, tensor fascia lata, iliopsoas, rectus femoris muscles

SECONDARY OUTCOMES:
VAS (Visual Analogue Scale) | 10 seconds for each session
  a psychometric scale that is generally used in pain scale surveys and this study participants will be asked to scale the uncomfortable feelings during the vibration

CONTACTS AND LOCATIONS:
Overall Officials: Ju Seok Ryu, M.D. PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Department of Rehabilitation Medicine, Seoul National University Bundang Hospital, Seoul National University College of Medicine, Seongnam-si, Gyeonggi-do, South Korea